CLINICAL TRIAL: NCT00861159
Title: Measurement Of RLIP76 Auto Antibodies in Human Serum In Adults With Rheumatologic Diseases.
Brief Title: RLIP76 in Human Serum in Adults With Rheumatologic Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to lack of staffing resources and subject interest
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Measurement of RLIP76 Auto Antibodies in Human Serum in Adults with Rheumatologic Disease., University of North Texas Health Science Center
Other Study IDs: 2008-31
Record Dates: First submitted 2008-09-29; First posted 2009-03-13 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Carotid Atherosclerosis
Keywords: RLIP76 Auto Antibodies
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
It is the investigators aim to determine the feasibility of directly detecting anti-RLIP76 auto-antibodies in human serum using prepared RLIP76 antigen peptides in persons with rheumatologic disease and persons without rheumatologic diesease ("healthy subjects").

DETAILED DESCRIPTION:
This is an exploratory study conducted to see the feasibility of measuring the anti-RLIP76 antibody and to standardize the methods for its measurement. We will perform these studies on blood samples obtained from human subjects after informed concent for blood draw for research purposes is obtained by the Clinical Research Co-ordinator (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+), non-pregnant subjects with previously diagnosed rheumatologic disease will be candidates for the study.

Exclusion Criteria:

* Children, pregnant women, prisoner, persons with any medical condition that precludes phlebotomy, and patients unwilling or unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The experimental populations subject to study will be 100 outpatients in the rheumatology clinic otherwise undergoing routinely scheduled phlebotomy for standard clinical care purposes.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
The focus of the present study is limited to establishing validated protocols for detection of anti-RLIP76 antibodies in human sera. | three years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Awasthi, MD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

REFERENCES:
- [Result] Margutti P, Matarrese P, Conti F, Colasanti T, Delunardo F, Capozzi A, Garofalo T, Profumo E, Rigano R, Siracusano A, Alessandri C, Salvati B, Valesini G, Malorni W, Sorice M, Ortona E. Autoantibodies to the C-terminal subunit of RLIP76 induce oxidative stress and endothelial cell apoptosis in immune-mediated vascular diseases and atherosclerosis. Blood. 2008 May 1;111(9):4559-70. doi: 10.1182/blood-2007-05-092825. Epub 2007 Nov 9. PMID 17993611
- [Result] Singhal SS, Yadav S, Singhal J, Zajac E, Awasthi YC, Awasthi S. Depletion of RLIP76 sensitizes lung cancer cells to doxorubicin. Biochem Pharmacol. 2005 Aug 1;70(3):481-8. doi: 10.1016/j.bcp.2005.05.005. PMID 15950949
- [Result] Huang X, Johansson SG, Zargari A, Nordvall SL. Allergen cross-reactivity between Pityrosporum orbiculare and Candida albicans. Allergy. 1995 Aug;50(8):648-56. doi: 10.1111/j.1398-9995.1995.tb02581.x. PMID 7503400
- [Result] Boyum A, Lovhaug D, Tresland L, Nordlie EM. Separation of leucocytes: improved cell purity by fine adjustments of gradient medium density and osmolality. Scand J Immunol. 1991 Dec;34(6):697-712. doi: 10.1111/j.1365-3083.1991.tb01594.x. PMID 1749920
- [Result] Bradford MM. A rapid and sensitive method for the quantitation of microgram quantities of protein utilizing the principle of protein-dye binding. Anal Biochem. 1976 May 7;72:248-54. doi: 10.1016/0003-2697(76)90527-3. No abstract available. PMID 942051
- [Result] Laemmli UK. Cleavage of structural proteins during the assembly of the head of bacteriophage T4. Nature. 1970 Aug 15;227(5259):680-5. doi: 10.1038/227680a0. No abstract available. PMID 5432063
- [Result] Towbin H, Staehelin T, Gordon J. Electrophoretic transfer of proteins from polyacrylamide gels to nitrocellulose sheets: procedure and some applications. Proc Natl Acad Sci U S A. 1979 Sep;76(9):4350-4. doi: 10.1073/pnas.76.9.4350. PMID 388439
- [Result] Stuckler D, Singhal J, Singhal SS, Yadav S, Awasthi YC, Awasthi S. RLIP76 transports vinorelbine and mediates drug resistance in non-small cell lung cancer. Cancer Res. 2005 Feb 1;65(3):991-8. PMID 15705900